CLINICAL TRIAL: NCT07235735
Title: The Effect of Laughter Yoga on Individual and Organizational Outcomes in Nurse Managers: A Longitudinal Study
Brief Title: The Effect of Laughter Yoga on Individual and Organizational Outcomes in Nurse Managers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, SERPİL SUBAŞI ÇAĞLAR, lecturer in the department of nursing management, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Laughter Yoga
Record Dates: First submitted 2025-09-19; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Burnout, Professional; Stress, Psychological; Compassion Fatigue; Quality of Life; Decision Making; Problem Solving; Work Performance
Keywords: Nurse Managers; Laughter Yoga; Burnout; Stress; Work-Life Balance; Decision Making; Problem Solving; Job Performance; Compassion Fatigue; Conflict Management; Organizational Outcomes; Professional Development
MeSH Terms: conditions — Burnout, Professional; Stress, Psychological; Compassion Fatigue; Burnout, Psychological | interventions — Laughter Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Laughter Yoga (Experimental): Structured group-based laughter yoga sessions, 2 times per week, 30-45 minutes each, for 8 weeks.
  Interventions: Behavioral: Laughter Yoga Program
- Control (No Intervention): Participants continue their routine work duties without any additional intervention.

INTERVENTIONS:
Behavioral: Laughter Yoga Program — This intervention consists of a structured Laughter Yoga Program designed for nurse managers. Each session includes breathing exercises, warm-up activities, guided and simulated laughter exercises (such as clapping, chanting, role-play laughter), and a short relaxation/meditation phase. Sessions are conducted in small groups by a certified facilitator. The program is delivered twice weekly for 8 weeks, with each session lasting approximately 30-45 minutes. The intervention is intended to reduce burnout, stress, and compassion fatigue, while improving decision-making, problem-solving, job performance, and work-life balance.
  Other Names: Laughter Therapy;; Laughter Exercises
  Arms: Experimental: Laughter Yoga

SUMMARY:
The goal of this clinical trial is to learn if laughter yoga can improve both individual and organizational outcomes in nurse managers. The main questions it aims to answer are:

* Does laughter yoga lower burnout and stress levels in nurse managers?
* Does laughter yoga improve work-life quality and job performance?
* Does laughter yoga help nurse managers make better decisions and solve problems more effectively?
* Does laughter yoga lower compassion fatigue and support positive approaches to workplace conflict? Researchers will compare a laughter yoga group with a control group to see if there are meaningful differences.

Participants will:

* Join structured laughter yoga sessions for a defined period (weekly sessions).
* Complete surveys before and after the program about stress, burnout, work-life quality, decision-making, problem solving, job performance, compassion fatigue, and conflict approaches.
* Continue their usual work while attending sessions.

DETAILED DESCRIPTION:
Nurse managers play a vital role in healthcare systems by ensuring the quality of nursing services, supporting staff, coordinating care, and solving organizational problems. However, the combination of administrative responsibilities, staff shortages, and high expectations often leads to stress, burnout, compassion fatigue, and difficulties in maintaining work-life balance. These conditions not only affect the individual health and well-being of nurse managers but also reduce team motivation, patient care quality, and overall organizational performance.

Laughter yoga is a mind-body practice that combines intentional laughter with breathing exercises. It does not rely on humor or jokes; instead, participants engage in guided group exercises that promote spontaneous and prolonged laughter. Scientific evidence suggests that laughter yoga can lower stress hormones, increase endorphins, improve mood, and strengthen social bonds. Although laughter yoga has been studied in various populations, there is a lack of randomized controlled trials (RCTs) specifically focusing on nurse managers and their professional challenges.

This randomized controlled trial aims to fill this gap by evaluating the individual and organizational outcomes of laughter yoga among nurse managers working in university and state hospitals.

The expected contribution of this study is to provide new evidence on a cost-effective, non-pharmacological intervention that can be easily integrated into hospital settings. If laughter yoga proves effective, it can be adopted as a sustainable strategy to support nurse managers' mental health, enhance their leadership capacity, and indirectly improve patient care and organizational outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Currently working as a nurse manager
* Having at least six months of managerial experience
* Continuing to serve as a nurse manager throughout the study period

Exclusion Criteria:

* Having previously received laughter yoga training
* Use of medications affecting general health components during the study (e.g., for depression, anxiety)
* Being pregnant
* Experiencing an acute stressful life event, such as the death of a close relative
* Having undergone abdominal surgery within the past 6 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-11 (Estimated); Primary Completion 2026-02-17 (Estimated); Study Completion 2026-03-17 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress (Perceived Stress Scale - PSS) | Baseline, 8 weeks, 3 months.
  Developed by Cohen & Williamson, adapted to Turkish by Eskin in 2013. 14 items, single-factor measure of stress.
  Scale Range: 0-56. Interpretation Higher scores = greater perceived stress (worse outcome).
Burnout Levels (Maslach Burnout Inventory - MBI) | Baseline, immediately post-intervention (8 weeks), and follow-up (3 months after intervention).
  Developed by Maslach & Jackson in 1986, adapted to Turkish by Ergin in1992. 22 items, three subscales: Emotional Exhaustion, Depersonalization, and Personal Accomplishment.
  Scale Range: Emotional Exhaustion (0-54), Depersonalization (0-30), Personal Accomplishment (0-48).
  Interpretation: Higher Emotional Exhaustion and Depersonalization scores = worse outcome; higher Personal Accomplishment scores = better outcome.

SECONDARY OUTCOMES:
Problem Solving Inventory | Baseline, 8 weeks, 3 months
  Problem Solving Inventory, Developed by Heppner & Peterson in1982; adapted to Turkish by Şahin in 1993
  Description: 31 items, six subscales: Problem-Solving Confidence, Approach-Avoidance, Personal Control, Planfulness, Impulsivity, Reflective Style.
  Scale Range: 31-186. Interpretation: Higher scores = less effective problem solving (worse outcome); lower scores = better problem-solving skills.
Work Performance | Baseline, 8 weeks, 3 months.
  Work Performance Job Performance Scale - Goodman and Svyantek in 1999; Turkish adaptation was made in 2014 by Bağcı.
  Description: 25 items, two subscales: Task Performance and Contextual Performance.
  Scale Range: 25-125. Interpretation: Higher scores = better work performance.
Compassion Fatigue | Baseline, 8 weeks, 3 months
  Developed by Dennis Portnoy and adapted Turkısh by Özdemir and Kutlu in 2022. The form consists of 40 items. The scale, which has no sub-dimensions, is evaluated based on the total number of items. The scale is a 3-point Likert-type scale: 1 = Very true, 2 = Partly true, and 3 = Rarely true. Those who answered "Very true" to 15 or more items in total are considered to have high levels of compassion fatigue.Cronbach alpha is 0,87
Decision-Making Styles scale | Baseline, 8 weeks, 3 months.
  Developed by Scott and Bruce in 1995; adapted to Turkish by Yılmaz Kuşaklı in 2023
  24 items, five subscales: Rational, Intuitive, Dependent, Avoidant, Spontaneous.
  Scale Range: 24-120. Interpretation: Higher scores in each subscale = more frequent use of that decision-making style

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Yang, Z., Huang, H., & Li, G. (2024). Status and influencing factors of work stress among nurse managers in western China: a cross-sectional survey study. BMC nursing, 23(1), 68. — https://scholar.google.com.tr/scholar?hl=tr&as_sdt=0%2C5&q=Status+and+influencing+factors+of+work+stress+among+nurse+managers%3A+A+cross-sectional+study+in+China&btnG=
- See also: Alici, N. K., & Dönmez, A. A. (2020). A systematic review of the effect of laughter yoga on physical function and psychosocial outcomes in older adults. Complementary therapies in clinical practice, 41, 101252. — https://scholar.google.com.tr/scholar?hl=tr&as_sdt=0%2C5&as_vis=1&q=The+effects+of+laughter+yoga+on+health-related+outcomes%3A+A+systematic+review.+Complementary+Therapies+in+Clinical+Practice&btnG=
- See also: Maslach, C., & Jackson, S. E. (1981). The measurement of experienced burnout. Journal of organizational behavior, 2(2), 99-113. — https://scholar.google.com/scholar?hl=tr&as_sdt=0%2C5&q=Maslach%2C+C.%2C+%26+Jackson%2C+S.+E.+%281981%29.+The+measurement+of+experienced+burnout.+Journal+of+organizational+behavior%2C+2%282%29%2C+99-113.&btnG=
- See also: Ergin, C. (1992). Doktor ve hemsirelerde tukenmislik ve Maslach tukenmislik olceginin uyarlanmasi. VII. Ulusal Psikoloji Kongresi, 22th September 1992 Ankara (Turkey). — https://cir.nii.ac.jp/crid/1570291225076829312
- See also: Bağcı, Z. (2014). ÇALIŞANLARIN İŞ DOYUMUNUN GÖREV VE BAĞLAMSAL PERFORMANSLARI ÜZERİNDEKİ ETKİSİ. Yönetim ve Ekonomi Araştırmaları Dergisi, 12(24), 58-72. — https://dergipark.org.tr/en/pub/yead/issue/21807/234392
- See also: UÇAR ÖZDEMİR, S., & KOCA KUTLU, A. (2022). Şefkat Yorgunluğu Ölçeği'nin Hemşireler Üzerinde Türkçe Geçerlilik ve Güvenilirliği Çalışması: Metodolojik Araştırma. Turkiye Klinikleri Journal of Nursing Sciences, 14(2). — https://www.turkiyeklinikleri.com/article/en-sefkat-yorgunlugu-olceginin-hemsireler-uzerinde-turkce-gecerlilik-ve-guvenilirligi-calismasi-metodolojik-arastirma-98273.html